CLINICAL TRIAL: NCT00359320
Title: A Randomized Trial of Two Surgical Techniques for Pancreaticojejunostomy in Patients Undergoing Pancreaticoduodenectomy
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Terminated by IRB
Sponsor: Thomas Jefferson University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 06U.198; JT 1258 (Other: JeffTrial Number); NCT00432848 (obsolete NCT alias)
Record Dates: First submitted 2006-08-01; First posted 2006-08-02 (Estimated); Last update posted 2025-05-02 (Actual); Status verified 2025-05

CONDITIONS: Pancreatic Neoplasms; Biliary Tract Neoplasms; Pancreatitis, Chronic; Duodenal Neoplasms
Keywords: Pancreaticoduodenectomy; Pancreaticojejunostomy; Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms; Biliary Tract Neoplasms; Pancreatitis, Chronic; Duodenal Neoplasms | interventions — Pancreaticojejunostomy

ARMS (1):
- Mucosa-to-jejunal mucosa technique of pancreaticojejunosto (Experimental): Determine whether a duct mucosa-to-jejunal mucosa technique of pancreaticojejunostomy will improve the pancreatic fistula rate
  Interventions: Procedure: pancreaticojejunostomy

INTERVENTIONS:
Procedure: pancreaticojejunostomy

SUMMARY:
The purpose of this trial is to determine whether a mucosa-to-mucosa technique of pancreaticojejunostomy will improve the pancreatic fistula rate.

DETAILED DESCRIPTION:
Pancreaticoduodenectomy (PD) is a commonly performed operative procedure which is used in selected patients with benign and malignant diseases of the pancreas and periampullary region. The procedure involves regional resection of the pancreatic head, neck, and uncinate process en-bloc with the duodenum, distal bile duct, and lymph nodes. The standard 'Whipple' operation also adds a distal gastrectomy to the above procedures, while a pylorus-preserving pancreaticoduodenectomy (PPPD) spares the distal stomach. The indications for PD include neoplastic processes confined to the periampullary region, such as pancreatic cancer, distal common bile duct cancer, duodenal cancer, ampullary cancer, neuroendocrine tumors, cystic tumors, etc. A small number of benign conditions, such as chronic pancreatitis and benign neoplasms are also treated with PD. Upon completion of the pancreatic resection, 3 anastomoses are used to re-establish GI continuity-a pancreatic-enteric anastomosis, a biliary-enteric anastomosis, and a gastro or duodeno-enteric anastomosis. The pancreatic-enteric anastomosis has traditionally been the most troubling of these anastomoses because of a failure to heal and resultant fistulas and leaks.

The operative mortality rate for PD is usually less than 5% in major surgical centers with significant experience with the procedure. The leading causes of mortality include hemorrhage, cardiac events, and sepsis (often related to a pancreatic-enteric fistula). In contrast to this low mortality rate, the morbidity rate is still quite high with one review showing a rate of 40%. One of the most common causes of morbidity is a leak or pancreatic fistula from the pancreatic-enteric anastomosis. A recent review estimated the incidence of this complication to be 10% to 28.5%. A pancreatic fistula is currently defined by the International Study Group for Pancreatic Fistulas (ISGPF) as drain amylase levels that are ≥3 times normal amylase levels from the third postoperative day onward, if drain output is ≥ 10ml, and if the color of the drained fluid is altered (non-serous). Several large single institution series from the Mannheim, Lahey, and Mayo Clinics have shown leak rates of 11-15%. The Mannheim Clinic series demonstrated that 20% of the pancreatic fistulas were directly responsible for postoperative deaths.

There have been several randomized prospective trials by investigators at the Johns Hopkins Hospital which have tested various interventions attempting to improve the leakage rates. In one trial, they determined that leak rates were similar (11-12%) whether the pancreatic-enteric anastomosis was a pancreaticojejunostomy (PJ) or a pancreaticogastrostomy (PG). In another trial, these investigators evaluated the use of prophylactic octreotide as an agent to reduce pancreatic fistula rates-in this study there was no decrease in fistula rates with the use of octreotide. Finally, these authors most recently performed a randomized, prospective trial of stenting the pancreatic-enteric anastomosis. In this trial, the fistula rates were not changed by the placement of a perioperative stent across the anastomosis.

There are two widely used methods for the PJ reconstruction after PD-invagination or 'dunking' the pancreatic remnant or end-to-side duct-to-mucosa PJ. In the invagination technique, the cut end of the pancreas in sewn into an opening in the side of the jejunum using two layers of suture-an outer layer of permanent suture on the pancreas capsule and bowel serosa and muscle, and an inner layer of running dissolvable suture on the duct and pancreatic parenchyma and full thickness of the bowel wall. In the duct-to-mucosa technique, there is again an outer layer of interrupted permanent suture. However, the inner layer is an interrupted anastomosis between the pancreatic duct and the bowel mucosa. In one single institution study utilizing the duct-to-mucosa technique and an internal stent, Strasberg et al demonstrated a pancreatic fistula rate of 1.6% in 123 patients. In another review by Tani et al, the fistula rate was 11% for the stented duct-to-mucosa technique and 6.5% for the 2 layer end-to-side externally stented technique.

There has been only one small randomized, prospective trial evaluating a duct-to-mucosa versus an end-to-side PJ reported in the literature. In this trial, the authors randomized 144 patients undergoing PD to either a 2-layer duct-to-mucosa anastomosis or a single layer end-to-side anastomosis which was not invaginated. Pancreatic fistulas were seen in 14% of patients-13% in the duct-to-mucosa group and 15% in the end-to-side group and there was no difference in complications between groups. It is not entirely clear from this study how these anastomoses were performed, but it does not appear that their construction was compatible to the methods that are most commonly used today.

Therefore, we propose to perform a randomized, prospective, controlled study comparing these two techniques. This study will be offered to all patients at Thomas Jefferson Hospital undergoing PD. Patients will be recruited on the basis of the preoperative anticipation of pancreaticoduodenal resection and preoperative consent will be obtained. Stratification and randomization will be performed intraoperatively, following pancreaticoduodenal resection. Because many studies have demonstrated that leak rates are directly related to pancreatic texture, we will stratify into two groups: soft (normal) texture (predicted fistula rate of 15-30%) and hard (fibrotic) texture (predicted fistula rate of 0-15%). Patients will be randomized to one of two groups: 1) pancreatic duct to jejunal mucosa, two-layer anastomosis or 2) end-to-side, two-layer, invagination technique.

The intraoperative management of the patients will not be influenced by this study and will be under the direction of the attending surgeon. The perioperative care of the patient, including the use of prophylactic antibiotics, gastric acid secretory inhibition agents, nasogastric tubes, the timing of removal of operatively placed closed-suction drains, and the restoration of oral intake will remain under the direction of the attending surgeon. If a postoperative pancreatic fistula does occur, the attending surgeon will manage the fistula appropriately. We have a Critical Pathway in place which we will use to standardize patient care and insure uniform postoperative management.

Immediately following the PD, the attending surgeon will complete a short questionnaire documenting the type of resection performed, the type of anastomosis, the character of the remnant pancreas, the size of the pancreatic duct, how the pancreas was transected (stapler, electrocautery, etc), and other details of the operative procedure. Other routine data that will be collected includes further details of the operative procedure (from the operative report), pathology of the resected specimen (from the pathology report), and occurrence of postoperative morbidity and mortality.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have undergone pancreaticoduodenectomy.
* Must have pancreatic remnant remaining in place (body and tail).
* Must be candidate for reconstruction by pancreaticojejunostomy by one of the two techniques described below.
* Must have an identifiable pancreatic duct which can be used for a duct-to-mucosa anastomosis.

Exclusion Criteria:

* Patients undergoing total pancreatectomy.
* Patients undergoing PD who have had previous left-sided pancreatic resection.
* Failure to sign informed consent.
* Failure to identify the pancreatic duct.
* Pregnant patients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2006-05-25 (Actual); Primary Completion 2008-07-12 (Actual); Study Completion 2008-07-12 (Actual)

PRIMARY OUTCOMES:
The primary endpoint will be the pancreatic fistula rate. | 1 year

SECONDARY OUTCOMES:
Length of hospitalization | 1 year
Percutaneous intervention rates | 1 year
Reoperation rates | 1 year
Morbidity | 1 year
Death | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Adam C Berger, MD, Principal Investigator — Thomas Jefferson University
Locations (1):
- Thomas Jefferson University Hospital, Philadelphia, Pennsylvania, United States

REFERENCES:
- [Derived] Berger AC, Howard TJ, Kennedy EP, Sauter PK, Bower-Cherry M, Dutkevitch S, Hyslop T, Schmidt CM, Rosato EL, Lavu H, Nakeeb A, Pitt HA, Lillemoe KD, Yeo CJ. Does type of pancreaticojejunostomy after pancreaticoduodenectomy decrease rate of pancreatic fistula? A randomized, prospective, dual-institution trial. J Am Coll Surg. 2009 May;208(5):738-47; discussion 747-9. doi: 10.1016/j.jamcollsurg.2008.12.031. PMID 19476827
- See also: Thomas Jefferson University Hospital — http://hospitals.jefferson.edu/